CLINICAL TRIAL: NCT03336866
Title: STAMPOUT: Study of Antibody for Methamphetamine Outpatient Therapy
Brief Title: Study of Antibody for Methamphetamine Outpatient Therapy
Acronym: STAMPOUT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InterveXion Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M200C-1801; U01DA045366 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-01

CONDITIONS: Methamphetamine-dependence; Methamphetamine Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo
- IXT-m200 (Experimental): Single 6 or 20 mg/kg intravenous dose of IXT-m200
  Interventions: Drug: IXT-m200

INTERVENTIONS:
Drug: Placebo — Normal saline
  Arms: Placebo
Drug: IXT-m200 — IXT-m200 is an anti-methamphetamine monoclonal antibody
  Other Names: ch-mAb7F9
  Arms: IXT-m200

SUMMARY:
This study evaluates the ability of IXT-m200 to change methamphetamine concentrations in blood and alter the way methamphetamine feels. Participants will receive either placebo, a low or high dose of IXT-m200, in addition to methamphetamine challenge doses.

DETAILED DESCRIPTION:
IXT-m200 is a monoclonal antibody that binds to methamphetamine in the blood. The main purpose of this study is to look at the effects of IXT-m200 on the pharmacokinetics of methamphetamine and on methamphetamine liking effects. Additionally, the study will determine IXT-m200 pharmacokinetics, safety and tolerability in subjects with methamphetamine use disorder. Qualified subjects will receive a single dose of IXT-m200 followed by up to 4 methamphetamine challenge doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an informed consent form.
* Subject must be able to verbalize understanding of the consent forms, provide written informed consent, and verbalize willingness to complete study procedures.
* Males or females between 21 to 50 years of age, inclusive. Female subjects should be of non-childbearing potential or, they should be nonpregnant, nonlactating, and agree to use medically acceptable forms of birth control from screening to end-of-study follow-up, or have a partner who has had a vasectomy. Male subjects need to have had a vasectomy or agree to use a condom and spermicide in addition to their female partners using a form of birth control. They should agree not to donate sperm for 90 days post IXT-m200 dose.
* Body mass index (BMI) between 18.0 and 35.0 kg/m2. Body weight ≥ 50 kg and ≤ 100 kg.
* Subjects have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, alanine aminotransferase, aspartate aminotransferase, and alkaline phosphatase) < 3 times the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 times the upper limit of normal.
* Subjects meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for METH use disorder and are not seeking treatment at the time of the study.
* Subjects will be experienced METH users with a history of non-therapeutic METH use for 2 or more years. Subjects must have experience with smoking or IV injection of METH.
* Current METH use (past 30 days) less than daily, self-reported and documented by calendar-based timeline follow-back.
* Primary current (past 30 days) route of METH self-administration other than IV (ie, smoking, snorting, or oral).
* Subjects agree not to take METH from any source outside of the study during their participation in the study. Subjects agree not to take substances that are structurally similar to METH.
* Subjects must provide a negative urine sample prior to admission to the unit on Day -1 for the study.

Exclusion Criteria:

* Subjects who have been treated with a monoclonal antibody (mAb) in the past year.
* Known or suspected allergy sensitivity to IXT-m200 based on known allergies to other mAbs.
* History of severe allergy (rash, hives, breathing difficulty, etc) to any medications.
* History of allergic or environmental bronchial asthma.
* Clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, GI, cardiovascular, pulmonary (including chronic asthma), endocrine (eg, diabetes), central nervous, or hematologic systems, or recent clinically significant surgery.
* Current diagnosis or history of major psychiatric illness in the past two years or other current psychiatric condition requiring medication, other than methamphetamine dependence.
* Considered by the PI to be at imminent risk of suicide or injury to self, others, or property, or the subject has attempted suicide with the past year. Past year history of, or current evidence for, suicidal ideation or those who were actively suicidal based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Current dependence on alcohol or heavy use defined as >28 alcoholic drinks per week if male and >21 drinks per week if female in last 30 days.
* Current dependence on other drugs except amphetamines, or marijuana and nicotine used in moderate amounts.
* History of seizure, epilepsy, severe head injury with residual neurologic effects, multiple sclerosis, or stroke.
* Abnormal pre-admission vital signs, physical examination, clinical laboratory, ECG, or any safety variable which is considered clinically significant for this population.
* History of cardiovascular disease.
* Treatment with any prescription medications or over the counter nutritional supplements within 14 days prior to the first dose of study medication.
* Ingestion of any approved prescription anti-obesity drug or taken any over-the-counter medication for weight loss within a period of 90 days prior to the first dose of study medication.
* Ingestion or use of any investigational medication or device within 30 days prior to the first dose of study medication.
* Acute illness within 5 days prior to the first dose of study medication, eg, flu syndrome, GI virus, or clinically significant indigestion (eg, reflux).
* Positive result for hepatitis B surface antigen (HBsAG), hepatitis C (HepC) antibody, hepatitis A immunoglobulin M (IgM), or HIV Viral Serology, or nucleic acid testing (NAT) tests at screening.
* Positive breath alcohol test or positive urine drug test for illicit substances on Day -1.
* Subjects with history of donated blood, plasma, or platelets in last 30 days, and who do not agree to refrain from blood, plasma, platelets, egg or sperm donation during the study period.
* Predominant or only route of METH self-administration is IV.
* Any subject judged by the PI or Sponsor (or designee) to be inappropriate for the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, MD, Principal Investigator — PRA Health Sciences; Peter Winkle, MD, Principal Investigator — Anaheim Clinical Trials
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, Anaheim, California
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Final datasets are expected to contain pharmacokinetic data on IXT-m200 and METH, subjective effects data, immunogenicity totals, and safety data. No individually identifiable private information will be distributed.
Time Frame: These datasets will be available for distribution following submission to the FDA of the Clinical Study Report and publication. They will be available for 2 years after the initial publication.
Access Criteria: These datasets and associated documentation will be made available on CD by the Sponsor to requestors under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology and not distributing to third parties; and (3) a commitment to destroying or returning the data after analyses are completed. Requests should be sent to intervexion@gmail.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two clinical research sites in Salt Lake City, UT and Anaheim, CA between April 2018 and October 2020.
Pre-assignment Details: Participants underwent drug discrimination testing on Day 1 (30 mg IV methamphetamine vs normal saline). Those who reported appropriate responses on drug effects questionnaires and had no safety concerns following IV methamphetamine dosing were allowed to continue in the study. 77 subjects were enrolled, 10 discontinued or withdrew after Day 1 and 11 did not pass drug discrimination and were disqualified.
Groups:
- IXT-m200, 6 mg/kg: Single 6 mg/kg intravenous dose of IXT-m200
  IXT-m200: IXT-m200 is an anti-methamphetamine monoclonal antibody
- IXT-m200, 20 mg/kg: Single IV dose of 20 mg/kg IXT-m200
Period: Overall Study
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Started | 20 | 18 | 18
Completed | 17 | 17 | 14
Not Completed | 3 | 1 | 4
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Noncompliance with clinic house rules | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- IXT-m200, 20 mg/kg: Single 20 mg/kg intravenous dose of IXT-m200
- Total: Total of all reporting groups
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg | Total
Number analyzed (Participants) | 20 | 18 | 18 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (7.34) | 32.2 (7.79) | 34.1 (7.40) | 33.7 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 10
  Male | 15 | 15 | 16 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 5
  Not Hispanic or Latino | 18 | 15 | 18 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 17 | 16 | 15 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 18 | 56
Weight [Mean (Standard Deviation); unit: kg] | 76.12 (13.109) | 75.15 (13.832) | 79.59 (12.624) | 76.92 (13.090)
Height [Mean (Standard Deviation); unit: cm] | 172.23 (10.827) | 171.32 (8.852) | 177.34 (7.093) | 173.58 (9.340)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.71 (3.953) | 25.56 (4.088) | 25.36 (4.056) | 25.55 (3.959)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Methamphetamine (METH) Area Under the Curve (AUCinf) Resulting From METH Challenge Doses Following Single IV Doses of IXT-m200
Description: METH AUCinf following IXT-m200 dosing on each METH Challenge Day.
Time Frame: Day 1, 5, 12, 19, and 26
Population: This outcome used the pharmacokinetic (PK) set. The PK set consisted of all subjects in the safety analysis set for whom at least 1 PK parameter could be calculated for METH or IXT-m200.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- IXT-m200, 6 mg/kg: Single 6 mg/kg intravenous dose of IXT-m200
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 18 | 18
h*ng/mL
  Day 1, AUCinf | 1635 (1345) | 1433 (555) | 1265 (350)
  Day 5, AUCinf: number analyzed (Participants) | 19 | 14 | 9
  Day 5, AUCinf | 1233 (323) | 14042 (3067) | 39379 (8288)
  Day 12, AUCinf: number analyzed (Participants) | 19 | 13 | 10
  Day 12, AUCinf | 1254 (341) | 8210 (2184) | 21846 (3915)
  Day 19, AUCinf: number analyzed (Participants) | 18 | 12 | 12
  Day 19, AUCinf | 1219 (346) | 5640 (1123) | 16458 (2580)
  Day 26, AUCinf: number analyzed (Participants) | 7 | 4 | 2
  Day 26, AUCinf | 1225 (389) | 4336 (1021) | 12411 (2597)
Statistical Analysis 1: Comparison: Placebo vs IXT-m200, 6 mg/kg; Values were compared by a statistical analysis of change from Day 1 in METH PK parameters following IXT-m200 dosing. Geometric LS Mean change from Day 1 for each treatment on each day were calculated. Geometric LS Means Ratios of change in METH exposure for each dose level of IXT-m200 compared to Placebo on each Day 5 (primary), Day 12, Day 19 and Day 26 were calculated along with the 95% confidence intervals; Test type: Other — The effect of IXT-m200 on METH exposure was evaluated with a linear mixed effects model. The response variable in the model was the natural-log transformed change in METH exposure parameters: AUCinf. The model contained fixed effects for treatment, day (categorical day postdose), natural-log transformed Day 1 baseline parameter and a treatment-by-day interaction, and a random effect for subject; p < 0.0001, Mixed Models Analysis — Geometric LS Means Ratios of change in METH exposure for IXT-m200 compared to Placebo on Day 5 (primary). Threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Geometric LS Means Ratios of change in METH exposure for IXT-m200 compared to Placebo on Day 12. Threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Geometric LS Means Ratios of change in METH exposure for IXT-m200 compared to Placebo on Day 19 (primary). Threshold for statistical significance was p<0.05
Statistical Analysis 4: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Geometric LS Means Ratios of change in METH exposure for IXT-m200 compared to Placebo on Day 26. Threshold for statistical significance was p<0.05
Statistical Analysis 5: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Geometric LS Means Ratios of change in METH exposure for IXT-m200 compared to Placebo on Day 19. Threshold for statistical significance was p<0.05
Statistical Analysis 8: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 4]

2. Primary Outcome: Change in Plasma Methamphetamine (METH) Maximum Concentration (Cmax) Resulting From METH Challenge Doses Following Single IV Doses of IXT-m200
Description: METH Cmax following IXT-m200 dosing on each METH Challenge Day.
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 18 | 18
ng/mL
  Day 1, Cmax | 111 (58) | 98 (29) | 90 (24)
  Day 5, Cmax: number analyzed (Participants) | 20 | 16 | 18
  Day 5, Cmax | 103 (56) | 312 (37) | 759 (135)
  Day 12, Cmax: number analyzed (Participants) | 20 | 16 | 16
  Day 12, Cmax | 100 (31) | 198 (24) | 444 (92)
  Day 19, Cmax: number analyzed (Participants) | 18 | 15 | 15
  Day 19, Cmax | 96 (36) | 168 (24) | 340 (57)
  Day 26, Cmax: number analyzed (Participants) | 7 | 5 | 3
  Day 26, Cmax | 80 (13) | 145 (17) | 262 (54)
Statistical Analysis 1: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — The effect of IXT-m200 on METH exposure was evaluated with a linear mixed effects model. The response variable in the model was the natural-log transformed change in METH exposure parameters: Cmax. The model contained fixed effects for treatment, day (categorical day postdose), natural-log transformed Day 1 baseline parameter and a treatment-by-day interaction, and a random effect for subject; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 4: Comparison: Placebo vs IXT-m200, 6 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs IXT-m200, 20 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 7]

3. Secondary Outcome: Change in Subjective Effects for CRAVE of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for CRAVE over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: The pharmacodynamic (PD) analysis set included 54 (96.4%) subjects for at least one time point. Two subjects were excluded after IXT-m200 dosing from the PD set due to having no measures for PD data due to early discontinuation. Other subjects were excluded for having no PD data at subsequent timepoints due to leaving the inpatient portion of the study early.
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 6601 (4492) | 7040 (6022) | 8658 (5133)
  Day 5 | 5758 (4642) | 5837 (5870) | 5980 (4363)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 4587 (4466) | 5544 (6318) | 5532 (3974)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 3456 (4406) | 6457 (6623) | 4426 (4292)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 3044 (3611) | 2374 (2683) | 5716 (9434)

4. Secondary Outcome: Change in Subjective Effects for DISLIKE of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for DISLIKE over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 2124 (2173) | 2806 (4517) | 1697 (2446)
  Day 5 | 2021 (2636) | 3331 (3966) | 2523 (3412)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 1998 (2598) | 3393 (5240) | 2292 (3176)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 2089 (2686) | 3433 (5486) | 2888 (4245)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 1610 (2434) | 1925 (3679) | 50520 (6042)

5. Secondary Outcome: Change in Subjective Effects for FEEL of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for FEEL over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 5963 (2731) | 10640 (4839) | 8116 (4242)
  Day 5 | 6470 (3886) | 9923 (5441) | 6822 (4089)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 5491 (4370) | 9179 (5318) | 7029 (4597)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 5827 (4723) | 10086 (5122) | 6078 (4772)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 5784 (3992) | 7405 (4315) | 9277 (7464)

6. Secondary Outcome: Change in Subjective Effects for GOOD of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for GOOD over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 6151 (2872) | 10984 (5214) | 8378 (3766)
  Day 5 | 6555 (4260) | 9783 (5185) | 6903 (3820)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 5584 (4498) | 9236 (5083) | 7001 (4211)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 6138 (5393) | 10016 (5209) | 5238 (3999)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 6335 (5099) | 7468 (3443) | 6760 (6967)

7. Secondary Outcome: Change in Subjective Effects for HIGH of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for HIGH over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 5873 (2671) | 10599 (4871) | 7947 (4218)
  Day 5 | 6187 (3744) | 9765 (5441) | 6813 (4046)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 5117 (4420) | 9162 (5245) | 6973 (4583)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 5494 (4916) | 9740 (5366) | 6018 (4700)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 5603 (3980) | 7562 (4542) | 9690 (7217)

8. Secondary Outcome: Change in Subjective Effects for LIKE of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for LIKE over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 7495 (3870) | 11322 (4276) | 9858 (3635)
  Day 5 | 7582 (4437) | 9668 (4997) | 7430 (4126)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 6394 (5089) | 9498 (5002) | 7111 (4001)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 6420 (5633) | 10271 (5432) | 6027 (3905)
  Day 26 | 7354 (5345) | 7713 (2827) | 6811 (7344)

9. Secondary Outcome: Change in Subjective Effects for MORE of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for MORE over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 9469 (4254) | 9404 (5347) | 11164 (4365)
  Day 5 | 8582 (4853) | 7341 (5671) | 7796 (4303)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 6629 (5306) | 7734 (6017) | 7802 (3954)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 5654 (5911) | 8521 (6584) | 5603 (4593)
  Day 26 | 6801 (6021) | 4059 (4201) | 5273 (8644)

10. Secondary Outcome: Change in Subjective Effects for STIMULATED of METH Challenge Doses
Description: Drug effects questionnaires (visual analog scales with range from 0 (no effect) to 100 (maximum effect)) were administered following weekly doses of methamphetamine starting on Day 5, one day after IXT-m200 or placebo administration. Participants were asked questions assessing subjective effects for STIMULATED over 180 minutes. Values were calculated as an area under the curve by using the trapezoidal rule; time 0 was set to 0 on the effect scale (at time of methamphetamine administration) and the area was calculated through 180 min post-dose. Lower values would indicate less drug effect (better) than higher values indicating larger drug effect (worse).
Time Frame: Day 1, 5, 12, 19, and 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale * min
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 16 | 18
score on a scale * min
  Day 1 | 6155 (3245) | 11041 (4934) | 8231 (4259)
  Day 5 | 6108 (3615) | 9902 (5445) | 6885 (3915)
  Day 12: number analyzed (Participants) | 20 | 16 | 16
  Day 12 | 5407 (4279) | 9502 (5234) | 6913 (4448)
  Day 19: number analyzed (Participants) | 18 | 15 | 15
  Day 19 | 5643 (4387) | 10314 (5130) | 5764 (4707)
  Day 26: number analyzed (Participants) | 7 | 5 | 3
  Day 26 | 5777 (3498) | 7062 (4436) | 9435 (7499)

11. Secondary Outcome: Safety and Tolerability of IXT-m200 Followed by METH Challenges
Description: Number of serious adverse events (SAEs) as identified by physical examinations and vital sign, adverse event, ECG, and clinical laboratory testing, and immune response by measurement of anti-IXT-m200 antibody levels.
Time Frame: 126 days
Population: All subjects who received a dose of IXT-m200 or placebo on Day 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 20 | 18 | 18
Participants | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetics of IXT-m200 Following Single Administration
Description: Measured by serum concentrations of IXT-m200 over time
Time Frame: 122 days
Population: All subjects who had quantifiable serum concentrations of IXT-m200 above the lower limit of quantitation (<1250 ng/mL) starting at the first time point within 2.25 hr post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IXT-m200, 6 mg/kg | IXT-m200, 20 mg/kg
Number analyzed (Participants) | 18 | 18
ng/mL
  Pre-dose | 617.1589 (2310.85995) | 101.9665 (432.60722)
  2.25 hr | 148344.5945 (36757.72368) | 437078.0551 (86546.28544)
  4 hr | 146618.9207 (31767.42539) | 413372.2737 (86725.33552)
  6 hr | 136095.9889 (38937.85634) | 399030.4857 (80456.98764)
  12 hr: number analyzed (Participants) | 17 | 18
  12 hr | 129181.7595 (34383.49379) | 357523.6776 (66912.58267)
  24 hr: number analyzed (Participants) | 16 | 18
  24 hr | 104920.1213 (16662.63925) | 308379.4673 (51024.44575)
  72 hr: number analyzed (Participants) | 16 | 18
  72 hr | 80955.9851 (14213.86691) | 261876.2091 (105541.51539)
  192 hr: number analyzed (Participants) | 16 | 16
  192 hr | 52338.2686 (10831.30591) | 165650.1889 (43060.62407)
  360 hr: number analyzed (Participants) | 16 | 15
  360 hr | 41457.508 (6880.32292) | 119773.4315 (26091.50216)
  528 hr: number analyzed (Participants) | 6 | 3
  528 hr | 30996.9615 (4340.51769) | 84460.7453 (12052.38197)
  576 hr: number analyzed (Participants) | 12 | 11
  576 hr | 28816.8833 (4801.42874) | 93827.4756 (28503.81089)
  744 hr: number analyzed (Participants) | 16 | 14
  744 hr | 22375.2957 (8092.25642) | 73363.3274 (22594.3438)
  912 hr: number analyzed (Participants) | 16 | 14
  912 hr | 16793.6838 (4465.29642) | 61311.3385 (20125.59405)
  1080 hr: number analyzed (Participants) | 17 | 13
  1080 hr | 12230.3541 (3819.65649) | 45940.3791 (12826.46281)
  1248 hr: number analyzed (Participants) | 17 | 13
  1248 hr | 10954.1343 (3596.63207) | 38972.226 (11834.15391)
  1416 hr: number analyzed (Participants) | 17 | 14
  1416 hr | 8321.6347 (2654.52136) | 29865.3018 (10122.90309)
  1920 hr: number analyzed (Participants) | 16 | 12
  1920 hr | 4493.8091 (2547.2715) | 16676.9182 (7385.34675)
  2424 hr: number analyzed (Participants) | 17 | 12
  2424 hr | 2093.7292 (1803.09651) | 10002.5426 (4197.70821)
  2928 hr: number analyzed (Participants) | 17 | 13
  2928 hr | 1128.2148 (1846.27013) | 5226.7547 (2209.49318)

ADVERSE EVENTS:
Time Frame: 126 days
Groups:
- All Subjects: Day 1-3: No Investigational Product administration; subjects were administered 30 mg METH and saline on Day 1 for drug discrimination.
- Placebo: Day 4-126: Normal saline
  Placebo: Normal saline
- IXT-m200, 6 mg/kg: Day 4-126: Single 6 mg/kg intravenous dose of IXT-m200
  IXT-m200: IXT-m200 is an anti-methamphetamine monoclonal antibody
- IXT-m200, 20 mg/kg: Day 4-126: Single 20 mg/kg intravenous dose of IXT-m200
Arm/Group | All Subjects: Day 1-3 | Placebo: Day 4-126 | IXT-m200, 6 mg/kg: Day 4-126 | IXT-m200, 20 mg/kg: Day 4-126
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/20 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/20 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 69/77 | 20/20 | 17/18 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects: Day 1-3 (N=77) | Placebo: Day 4-126 (N=20) | IXT-m200, 6 mg/kg: Day 4-126 (N=18) | IXT-m200, 20 mg/kg: Day 4-126 (N=18)
Palpitations (Cardiac disorders) | 14 | 8 | 7 | 8
Tachycardia (Cardiac disorders) | 7 | 3 | 8 | 5
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pruritis (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Eye irritation (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Scleral haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Scleral disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vision blurred (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Visual impairment (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 8 | 5 | 3 | 3
Nausea (Gastrointestinal disorders) | 4 | 4 | 2 | 5
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal distension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Submaxillary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 10 | 4 | 5 | 6
Catheter site pain (General disorders) | 3 | 5 | 2 | 3
Feeling hot (General disorders) | 15 | 4 | 3 | 3
Influenza like illness (General disorders) | 0 | 3 | 2 | 2
Fatigue (General disorders) | 4 | 3 | 2 | 0
Feeling abnormal (General disorders) | 4 | 2 | 1 | 1
Energy increased (General disorders) | 6 | 1 | 2 | 0
Chills (General disorders) | 0 | 2 | 0 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 1 | 1
Infusion site pain (General disorders) | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1
Catheter site nodule (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Medical device site reaction (General disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 1 | 3 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 11 | 6 | 6
Paraesthesia (Nervous system disorders) | 5 | 1 | 6 | 0
Dizziness (Nervous system disorders) | 7 | 1 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Vibratory sense increased (Nervous system disorders) | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 37 | 16 | 15 | 13
Hypervigilance (Psychiatric disorders) | 20 | 10 | 10 | 6
Anxiety (Psychiatric disorders) | 2 | 1 | 2 | 0
Bruxism (Psychiatric disorders) | 6 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0
Logorrhoea (Psychiatric disorders) | 3 | 1 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anhedonia (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Disinhibition (Psychiatric disorders) | 0 | 0 | 1 | 0
Disturbance in sexual arousal (Psychiatric disorders) | 2 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 4 | 0 | 0 | 1
Sleep terror (Psychiatric disorders) | 0 | 0 | 1 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 5 | 7 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Blister rupture (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Drug abuser (Social circumstances) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Disgeusia (Nervous system disorders) | 2 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0
Change in sustained attention (Psychiatric disorders) | 1 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 3 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
All participants were dosed with methamphetamine on a weekly basis following treatment with IXT-m200 or placebo. Thus, safety of IXT-m200 alone cannot be distinguished from the expected adverse events resulting from the methamphetamine doses. Variability of the responses on the drug effects questionnaires was much higher than anticipated. This resulted in insufficient power to detect differences between treated and control groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor agrees that the Investigator may present and publish methods and results of the study, but only after Sponsor has first published the results and with Sponsor's written permission. PRA shall provide to Sponsor any proposed presentation or publication for review 30 days prior to submission so that Sponsor may review for accuracy and provide comments and/or remove its proprietary or confidential information. PRA agrees that all reasonable comments will be incorporated.

DOCUMENTS (3):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03336866/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03336866/SAP_002.pdf
  • Informed Consent Form (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03336866/ICF_000.pdf